CLINICAL TRIAL: NCT04773171
Title: Efficacy of Computer-assisted Cognitive Remediation in Patients With Schizophrenia: A Randomized Controlled Trial
Brief Title: Efficacy of Computer-assisted Cognitive Remediation in Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HongKongPUDA
Record Dates: First submitted 2021-02-08; First posted 2021-02-26 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Schizophrenia; Psychosis; Cognitive Impairment; Executive Function; Randomized Controlled Trial; Efficacy
Keywords: Randomized Controlled Trial; Computer-assisted Cognitive Remediation; Executive Function
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CACR Group (Experimental): Participants of CACR group will attend individual computer-assisted cognitive remediation sessions. Researcher will give instruction in the use of the computerized training programs and assists participants during their training sessions.
  Interventions: Other: Computer-assisted Cognitive Remediation
- TAU Group (Active Comparator): Participants of TAU group will attend usual training sessions offered by the training centres with similar intensity and frequency as the CACR training.
  Interventions: Other: Conventional training programmes

INTERVENTIONS:
Other: Computer-assisted Cognitive Remediation — Drill practice and bridging activities
  Arms: CACR Group
Other: Conventional training programmes — Existing conventional activities in the settings
  Arms: TAU Group

SUMMARY:
Objective: To determine the efficacy of computer-assisted cognitive remediation (CACR) in patients with chronic schizophrenia in the community settings.

Study Design: Single-blinded prospective, pre-test/post-test randomized controlled trial (RCT) will be conducted in 2 groups of participants that receiving training in community settings. Treatment groups will attend individualized CACR programme using CogniPlus® while control group will continue attend conventional treatment as usual (TAU). Assessment on the means difference in assessing functions will be done after the study.

Samples: 80 patients with stable and chronic schizophrenia will be recruited from the community, using a sampling frame of selected diagnosis and homogeneity.

Expected Findings: Find out the training effects of selected CACR on EF and daily functioning in patients with schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is one of the most serious and disabling mental disorders. Prevalence of schizophrenia is about 1% worldwide. The related dysfunctions have great impact and burden to the concerned person and to the society. With increasing use of CR programmes in helping the patients to resume their capability in community living, the clinical outcome was not fully established especially on specific cognitive domains such as executive function (EF). The present study aims at evaluating the efficacy of CACR on developing EF and improving daily functioning. The result will provide information for therapists' future clinical decisions for patients' best reintegration into the societies. This also helps decrease the burden of family, society in the long run.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia, based on Diagnostic and statistical manual of mental disorders (5th ed.), at chronic and stable state
* Age from 18 to 64
* Regular attendance to rehabilitation training programmes
* Willing and capable to participate and are voluntarily consent to the participation
* Pass the cut-off point of referenced screening tests

Exclusion Criteria:

* Comorbid differential diagnosis
* History of organic brain disorder
* Complicated conditions that preclude regular attendance of the training
* Currently receiving computer-assisted cognitive remediation and other individual intensive cognitive training

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Change of Wisconsin Card Sorting Test Score | Baseline, after completion of half of the programme (an average of 6 weeks), one month post-treatment
  It is a neuropsychological test that is used to measure high-level cognitive processes as attention, perseverance, working memory, abstract thinking, cognitive flexibility, and set shifting.
  The test consists of 128 card designs, participant is required to sort the cards under the categorization rules and feedback from examiner in about 20 minutes. The more categories achieved (range 0 to 6) and less perseverative errors (out of 128 trials) the better executive control. Moreover, the lower the total number of trials administered (total number of cards used) reflects greater efficiency of the participant in the task; in addition, the greater the total number of correct responses (number of successes in combinations according to the category) and the lower the total number of errors (number of incorrect combinations) also indicate the better the participant's performance.
Change of The Digit Span Test Score (Digit Span Forward and Digit Span Backward) | Baseline, after completion of half of the programme (an average of 6 weeks), one month post-treatment
  It measures a participant's attention and working memory. Forward span captures attention capacity and backward span reflects working memory. The higher both the scores the better functioning. Participant repeats or reverses the digit sequencing after the examiner read out lists of random numbers, extra digit would be added for increased level of difficulty with two trials per level until the participant gives out incorrect answer. Average adult score for forward span is eight to ten and seven to nine for backward span.
Change of Cognitive scores in the cognitive remediation programme CogniPlus® | Through study completion, an average of 12 weeks
  There are 15 individual training modules that grouped into 6 function dimensions (attention, neglect/visual field training, memory, executive function, spatial processing and visuomotor skills) in this programme.
  Different number of difficulty levels and specific requirements are structured in different modules. For example, DATEUP module in memory dimension contains 25 levels, incremented with increasing number of stimuli that move in higher speed for the participants to retain and update the information; while ALERT module in attention dimension have 18 difficulty levels, with decreasing maximum permitted reaction time for the participants to respond.
  For the evaluations of results in all modules, the higher percentage of correct response, the shorter reaction/working time and the higher difficulty level attained indicate the better corresponding functioning. The importance of these cognitive scores is to help tracking the participants' task functioning throughout the study.
Change of Role Functioning Scale | Baseline, after completion of half of the programme (an average of 6 weeks), one month post-treatment
  It is a measure of functioning level of adults in four domains: working productivity, independent living/self-care, immediate social network relationships and extended social network relationships.
  7-point scale for the four domains and their total score (ranging from 4 to 28) represent the Global Role Functioning Index, the higher scores the better the person's functioning.

CONTACTS AND LOCATIONS:
Overall Officials: David Man, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- New Life Psychiatric Rehabilitation Association, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No